CLINICAL TRIAL: NCT05286944
Title: Mobile Phone Daily Alarm To Improve Compliance Of Intranasal Corticosteroid Among Allergic Rhinitis Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: UKM PPI/111/8/JEP-2019-819
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2021-03

CONDITIONS: Rhinitis, Allergic; Compliance, Medication
Keywords: allergic rhinitis; Intranasal steroid spray; compliance; mobile alarm
MeSH Terms: conditions — Rhinitis, Allergic; Medication Adherence; Patient Compliance

STUDY DESIGN:
Intervention Model Description: Single blinded randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant will be assigned a study number based on the recruitment timeline and assigned into the pre-randomized groups. Throughout the study, the primary investigator will not know which group is assigned for the mobile phone daily alarm. A second investigator will select the group for mobile phone daily alarm and set the alarm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile daily alarm (Experimental): A mobile smartphone with functioning alarm system and solely owned by the patient. The alarm will be set by the second investigator to alert the participant between 6am - 10am (based on participant's preference) in the morning daily. A recorded dual-language (English and Malay version) tone for alarm mobile phone will be used. Apart from that participants are also counseled and educated about allergic rhinitis and are also asked to fill up self monitored adherence card to document their nasal steroid intake.
  Interventions: Other: Mobile phone alarm reminder
- Control (No Intervention): This group of participant will receive counseling and education regarding allergic rhinitis and the importance of compliance. Patients are also given a self monitored adherence card to document their nasal steroid intake.

INTERVENTIONS:
Other: Mobile phone alarm reminder — Patients are reminded to take their INCS using a mobile phone alarm set to ring daily
  Arms: Mobile daily alarm

SUMMARY:
This is a randomized controlled trial to compare the compliance of allergic rhinitis patients towards intranasal steroids between those who use mobile daily alarm reminder and those who do not.

DETAILED DESCRIPTION:
In this single blinded RCT, adults with allergic rhinitis are randomized into either he intervention or control arm. The intervention involves installing an alarm with a prerecorded nmessage "Have you take your intranasal steroids" which will automatically ring every day on the patients mobile phone. The control arm do not have any alarm set up. Both groups are offered counseling and education regarding the importance of compliance to intranasal steroid upon recruitment. Daily reminder to take medication may eliminate reason for forgetting medication schedule, hence, improve compliance towards INCS among patients with allergic rhinitis. This study aims to assess the effectiveness of using daily mobile alarm on patient's compliance towards INCS.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 15 years old to 60 years old with persistent AR

  * Positive SPT towards DF, DP, BT, cockroach, Aspergillus, Cat fur
  * Own and able to operate functioning mobile smartphone with built in alarm
  * Able to understand simple instructions
  * Patients who can read in English and Malay
  * Newly diagnosed AR or previous patients who only take intranasal corticosteroid less than 4 times per week

Exclusion Criteria:

* • Patients on immunotherapy

  * Patients with mild intermittent AR
  * Pregnant patients
  * Patient with psychiatric illness
  * Patients with gross anatomical obstruction (severe DNS, gross polyposis, nasal tumour)
  * Chronic rhinosinusitis(CRS) with or without nasal polyposis
  * Patients who have adverse reaction towards INCS
  * Patients with severe hearing loss

Ages: 15 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2020-01-19 (Actual); Primary Completion 2022-06-22 (Estimated); Study Completion 2022-06-22 (Estimated)

PRIMARY OUTCOMES:
Compliance | 30 days
  Compliance was taken as 2/3rd use of INCS (20 days out of 30) = 20 x 0.38 = 7.6 g reduced weight.

CONTACTS AND LOCATIONS:
Overall Officials: Aneeza K W Hamizan, MD, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Universiti Kebangsaan Malaysia Medical center, Kuala Lumpur, WP Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katelaris CH, Lai CK, Rhee CS, Lee SH, Yun WD, Lim-Varona L, Quang VT, Hwang J, Singh H, Kim J, Boyle JM, Dhong HJ, Narayanan P, Vicente G, Blaiss M, Sacks R. Nasal allergies in the Asian-Pacific population: results from the Allergies in Asia-Pacific Survey. Am J Rhinol Allergy. 2011 Sep-Oct;25 Suppl 1:S3-15. doi: 10.2500/ajra.2011.25.3674. PMID 22185687
- [Background] Ho TM, Murad S, Kesavapillai R, Singaram SP. Prevalence of allergy to some inhalants among rhinitis patients in Malaysia. Asian Pac J Allergy Immunol. 1995 Jun;13(1):11-6. PMID 7488338
- [Background] Yuen AP, Cheung S, Tang KC, Ho WK, Wong BY, Cheung AC, Ho AC. The skin prick test results of 977 patients suffering from chronic rhinitis in Hong Kong. Hong Kong Med J. 2007 Apr;13(2):131-6. PMID 17406040
- [Background] Stanaland BE. Once-daily budesonide aqueous nasal spray for allergic rhinitis: a review. Clin Ther. 2004 Apr;26(4):473-92. doi: 10.1016/s0149-2918(04)90050-1. PMID 15189745
- [Background] Bridgeman MB. Overcoming barriers to intranasal corticosteroid use in patients with uncontrolled allergic rhinitis. Integr Pharm Res Pract. 2017 May 4;6:109-119. doi: 10.2147/IPRP.S129544. eCollection 2017. PMID 29354557
- [Background] Trangsrud AJ, Whitaker AL, Small RE. Intranasal corticosteroids for allergic rhinitis. Pharmacotherapy. 2002 Nov;22(11):1458-67. doi: 10.1592/phco.22.16.1458.33692. PMID 12432972
- [Background] Wong GW, Leung TF, Ko FW. Changing prevalence of allergic diseases in the Asia-pacific region. Allergy Asthma Immunol Res. 2013 Sep;5(5):251-7. doi: 10.4168/aair.2013.5.5.251. Epub 2013 Mar 18. PMID 24003381
- [Background] Jansen A, Andersen KF, Bruning H. Evaluation of a compliance device in a subgroup of adult patients receiving specific immunotherapy with grass allergen tablets (GRAZAX) in a randomized, open-label, controlled study: an a priori subgroup analysis. Clin Ther. 2009 Feb;31(2):321-7. doi: 10.1016/j.clinthera.2009.02.005. PMID 19302904
- [Background] Marple BF, Fornadley JA, Patel AA, Fineman SM, Fromer L, Krouse JH, Lanier BQ, Penna P; American Academy of Otolaryngic Allergy Working Group on Allergic Rhinitis. Keys to successful management of patients with allergic rhinitis: focus on patient confidence, compliance, and satisfaction. Otolaryngol Head Neck Surg. 2007 Jun;136(6 Suppl):S107-24. doi: 10.1016/j.otohns.2007.02.031. PMID 17512862
- [Background] Loh CY, Chao SS, Chan YH, Wang DY. A clinical survey on compliance in the treatment of rhinitis using nasal steroids. Allergy. 2004 Nov;59(11):1168-72. doi: 10.1111/j.1398-9995.2004.00554.x. PMID 15461597
- [Background] Braido F, Baiardini I, Puggioni F, Garuti S, Pawankar R, Walter Canonica G. Rhinitis: adherence to treatment and new technologies. Curr Opin Allergy Clin Immunol. 2017 Feb;17(1):23-27. doi: 10.1097/ACI.0000000000000331. PMID 27875376
- [Background] Wittig-Wells D, Higgins M, Carter J, Davis E, Holmes E, Jacob A, Samms-McPherson J, Simms S. Impact of a Preset Daily Cell Phone Alarm on Medication Adherence for Aspirin as Antithrombotic Therapy. Orthop Nurs. 2019 Sep/Oct;38(5):311-316. doi: 10.1097/NOR.0000000000000592. PMID 31568119
- [Background] Bousquet J, Van Cauwenberge P, Khaltaev N; Aria Workshop Group; World Health Organization. Allergic rhinitis and its impact on asthma. J Allergy Clin Immunol. 2001 Nov;108(5 Suppl):S147-334. doi: 10.1067/mai.2001.118891. No abstract available. PMID 11707753
- [Background] Wan Ishlah L, Gendeh BS. Skin prick test reactivity to common airborne pollens and molds in allergic rhinitis patients. Med J Malaysia. 2005 Jun;60(2):194-200. PMID 16114160
- [Result] Pizzulli A, Perna S, Florack J, Pizzulli A, Giordani P, Tripodi S, Pelosi S, Matricardi PM. The impact of telemonitoring on adherence to nasal corticosteroid treatment in children with seasonal allergic rhinoconjunctivitis. Clin Exp Allergy. 2014 Oct;44(10):1246-54. doi: 10.1111/cea.12386. PMID 25109375
- See also: Reference — http://www.researchgate.net/publication/325990822_Chinese_Society_of_Allergy_Guidelines_for_Diagnosis_and_Treatment_of_Allergic_Rhinitis